CLINICAL TRIAL: NCT05149040
Title: Very Elderly Patients' Treatment Preferences and Participation in Shared Decision-making in the Event of Acute Life-threatening Illness
Brief Title: Intensive Care of Elderly: What do They Wish for Themselves?
Status: Active, not recruiting | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor
Other Study IDs: 277504
Record Dates: First submitted 2021-10-31; First posted 2021-12-08 (Actual); Results first posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2024-12

CONDITIONS: Aged, 80 and Over; Critical Illness
Keywords: consent; goals of treatment; proxy accuracy; shared decision making
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- very elderly outpatients: outpatients (eyes, ear-nose-and throat, orthopaedic outpatient clinics at Haukeland University Hospital, Bergen, Norway) aged 80 years and older
  Interventions: Other: survey "Intensive care of very elderly: What do they wish for themselves?"
- proxy: next of kin who likely would act as a proxy in a medical emergency, identified by the very elderly respondent
  Interventions: Other: survey "Intensive care of very elderly: What do they wish for themselves?"

INTERVENTIONS:
Other: survey "Intensive care of very elderly: What do they wish for themselves?" — self-administered mailed survey

SUMMARY:
Do very elderly adults wish intensive care in the event of acute life-threatening illness and are their next of kin able to predict these preferences?

Very elderly patients are a steeply increasing patient population in intensive care units (ICUs), but the overall benefit of intensive care for these patients remains controversial. Will ICU admission improve survival and quality of life, or will it prolong suffering and delay natural death? Little is known about very elderly Norwegians life sustaining treatment (LST) preferences in these situations where treatment benefit is uncertain.

This project aims to improve critically ill very elderly patients' ICU trajectories by bringing forth knowledge about their treatment preferences, their family members' ability to predict these preferences, and by directing attention to the challenges of consent to critical care in cases of medical uncertainty.

A selv administered, mailed survey will be distributed among 400 outpatients aged 80 years or older and their next of kin. Respondents will be recruited at the ophthalmologic, ear-nose-and-throat and orthopaedic outpatient clinics at Haukeland University Hospital Bergen, Norway.

The investigators developed and validated a survey tool for this purpose, containing 3 hypothetical scenarios of acute life-threatening illness. The scenarios are randomly chosen from 20 hypothetical patient histories and are representative for ICU admission diagnoses in Norway and Europe. The participants will be asked for treatment choices, i.e. wishing admission to intensive care or not. A response option 'not wishing to engage in the treatment decision' is also provided.

Furthermore, the questionnaire includes factors that may influence elderlies' treatment preferences and proxies' ability to predict these preferences including: demographics, religion, previous experience with and / or communication about critical illness, comorbidity, frailty, quality of life, and projections (i.e. the proxy's own treatment preferences).

The respondents are requested to explain their choices by free-text comments after each scenario. They are also asked to elaborate how they wish next-of-kin should contribute to decision making in these cases. Additional space for free-text comments is provided in the end of the questionnaire.

The study design is exploratory. Responses will be analysed with both quantitative statistics and qualitative methods.

ELIGIBILITY:
Inclusion Criteria: Outpatients aged 80 years or older who register for appointment at the ophthalmologic, ear-nose-and-throat, and orthopaedic outpatient clinic at Haukeland University Hospital, Bergen, Norway.

Exclusion Criteria:

1. not consenting to participate
2. living in permanent care facility / nursing home
3. not able to complete the questionnaire owing to:

   * severely reduced vision / blindness
   * high degree of frailty (Clinical frailty scale ≥ 7)
   * cognitive impairment

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Community dwelling very elderly outpatients in the catchment area of Haukeland University Hospital, i.e. Greater Bergen Region, Western Norway.
Sampling Method: Non-Probability Sample
Enrollment: 1472 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2025-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Leonie I Schwarz, MD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1043 very old outpatients were approached. The next-of-kin respondents were recruited by the enrolled very old respondents.
Period: Overall Study
Arm/Group | Very Elderly Outpatients | Proxy
Started | 736 | 736
Completed | 202 | 153
Not Completed | 534 | 583

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Very Elderly Outpatients | Proxy | Total
Number analyzed (Participants) | 202 | 153 | 355
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age, Continuous (very old outpatients) | 86 (3.9) | 66 (13.3) | 82.8 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 116 | 218
  Male | 100 | 37 | 137
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Older Respondents Treatment Preferences in an Event of Acute Life-threatening Illness Warranting ICU Admission as Stated by Themselves and by Their Next of Kin Acting as Proxy
Description: Three mutually exclusive answer options in three randomly assigned clinically scenarios of acute critical illness in advanced age
  1. Wishing ICU admission
  2. Not wishing ICU admission
  3. Not wanting to decide
Time Frame: within 2 weeks of recruitment / upon completion of the questionnaire
Measure: Count of Units; unit: Treatment preference statement
Units Other Than Participants: Treatment preference statement
Arm/Group | Very Elderly Outpatients | Proxy
Number analyzed (Participants) | 202 | 153
Number analyzed (Treatment preference statement) | 590 | 453
Treatment preference statement
  Wishing ICU admission | 228 | 231
  Not wishing ICU admission | 238 | 154
  Not wanting to decide | 124 | 68

ADVERSE EVENTS:
Time Frame: 2 months
Description: Participants were offered to connect by phone or e-mail in the event of discomfort or distress during survey completion.
  All-Cause Mortality and Serious Adverse Events were not monitored.
Arm/Group | Proxy | Very Elderly Outpatients
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/202 | 0/153

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-06): https://cdn.clinicaltrials.gov/large-docs/40/NCT05149040/Prot_SAP_000.pdf